CLINICAL TRIAL: NCT01887392
Title: The Evaluation of a Multifaceted, Knowledge Translation Education Intervention in Long-Term Care and Its Ability to Facilitate the Uptake of Osteoporosis Canada 2010 Clinical Practice Guidelines, Across Ontario LTC Homes
Brief Title: Gaining Optimal Osteoporosis Assessments in Long-Term Care (GOAL)
Acronym: GOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Hamilton Health Sciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REB 13-229
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2016-12

CONDITIONS: Osteoporosis
Keywords: Long-term Care; Knowledge Translation
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wave A (Experimental): LTC Homes randomized into Wave A will receive the intervention first. The intervention includes Knowledge Translation Education Sessions.
  Interventions: Other: Knowledge Translation Education Sessions
- Wave B (Experimental): LTC Homes randomized into Wave B will receive the intervention after Wave A. The intervention includes Knowledge Translation Education Sessions.
  Interventions: Other: Knowledge Translation Education Sessions

INTERVENTIONS:
Other: Knowledge Translation Education Sessions — Two interactive sessions will be delivered to the interprofessional team at Month 1 and Month 6 and are 1 hour in length. The Clinical Consultant Pharmacist at each LTC home will lead the Knowledge Translation Sessions. Participants will watch an educational video, developed by the co-investigators with expertise in osteoporosis and geriatrics and members of the Ontario College of Family Physicians. Accompanying materials that support the topics in the video will be provided. Following the educational video, one of the experts from the video will phone the LTC home to address questions and provide the home with direct access to an expert.

SUMMARY:
The aim of this study is to disseminate the 2010 Osteoporosis Canada clinical practice guidelines, using a multi-faceted Knowledge Translation (KT) model, as KT aims to close the gap between knowledge generated from research and practice. The investigators' primary objective is to evaluate if this intervention can increase the percent of long-term care (LTC) residents receiving appropriate treatment for osteoporosis (i.e. treatment is considered appropriate for an individual over age 50 who has had a diagnosis of osteoporosis or a fragility fracture of the hip or vertebrae and those who have had more than one fragility fracture and is therefore considered high-risk). A secondary objective is to examine whether the intervention increases the percent of all LTC residents receiving Vitamin D equivalent to ≥800 IU/day.

DETAILED DESCRIPTION:
Individuals who live in LTC are at high risk for osteoporosis and fractures, particularly hip fractures, which lead to pain and transfer to acute care. The investigators' previous work in LTC has shown that awareness and use of clinical practice guidelines in LTC are low. To successfully transfer knowledge, it is imperative to understand the needs of the LTC teams and to tailor KT interventions appropriately.

Interventions which focus on strategies to overcome barriers and on new ways to deliver and promote the uptake of best practices that are specific to both the learning needs of LTC health care providers and the operational/organizational culture in LTC are greatly needed. Interdisciplinary teams who participated in the Vitamin D and Osteoporosis Study (ViDOS) indicated several process barriers that may hinder the proper identification and treatment of fractures in LTC. There is a need to educate Ontario LTC practitioners on the osteoporosis guidelines. The investigators' aim is to facilitate the uptake of Osteoporosis Canada 2010 Clinical Practice Guidelines, across Ontario LTC homes using the ViDOS multi-faceted KT model. Furthermore, the investigators will have a greater emphasis on the implementation of guidelines which includes risk assessment and appropriate medication use.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 2 physicians for each LTC home served by a Pharmacy provider

Exclusion Criteria:

* LTC homes that have only one prescribing physician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6800 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Difference in the percentage of residents appropriately prescribed an osteoporosis medication before and after the intervention. | 18 months
  Difference in the percentage of residents appropriately prescribed an osteoporosis medication before and after the intervention will be measured. Medications to be included in the baseline and post data download are in accordance with the current Osteoporosis Canada guidelines. Treatment is considered appropriate for an individual over age 50 who has had a diagnosis of osteoporosis or a fragility fracture of the hip or vertebra and those who have had more than one fragility fracture (i.e. high risk).

SECONDARY OUTCOMES:
Difference in the percentage of residents prescribed Vitamin D (equivalent to ≥800 IU/day) before and after the intervention. | 18 months
  Vitamin D will be included in the baseline and post data download to compare the two results and see if more residents have been prescribed vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- St. Peter's Hospital, Hamilton, Ontario, Canada